CLINICAL TRIAL: NCT06836700
Title: Comparison of Trifecta Analysis of Standard Versus Mini Percutaneous Nephrolithotomy in the Management of Urolithiasis
Acronym: Trifecta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hayat Abad Medical Complex, Peshawar (Other Government)
Responsible Party: Principal Investigator, Abdul Haseeb, Post Graduate Resident, Hayat Abad Medical Complex, Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 341/Chairman/R&E/Comittee; Institute of Kidney Diseases (Other: Institute of Kidney Diseases)
Record Dates: First submitted 2025-02-11; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Renal Stones; Urolithiasis, Calcium Oxalate
Keywords: Renal stone; PCNL
MeSH Terms: conditions — Nephrolithiasis; Nephrolithiasis, Calcium Oxalate

STUDY DESIGN:
Intervention Model Description: This study was executed as a single institution prospective cohort study at the department of urology, Institute of Kidney Diseases, Peshawar, Pakistan. The study was conducted between January 2022 and March 2024, focusing on patients who were eligible for percutaneous nephrolithotomy (PCNL) for stone treatment.
  After getting IREB approval from the Institute of Kidney Diseases, Peshawar, (certificate no 341), all participants received a detailed explanation of the study objectives, methodology, potential benefits, and risks before providing informed consent.
  Sample Size Calculation & Patient Selection:
  The sample size was determined using OpenEpi calculator and a total of 180 consecutive patients scheduled for PCNL were selected from an initial sample frame of 200. To maintain randomness in group allocation, a simple random sampling technique using the lottery method was applied. Patients were equally distributed into two Groups:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mini PCNL Group (Active Comparator): Participant in this group were subjected to MINI PCNL procedure.
  Interventions: Procedure: Mini PCNL
- Standard PCNL Group (Active Comparator): Participants in this group were subjected to Standard PCNL procedure
  Interventions: Procedure: Mini PCNL

INTERVENTIONS:
Procedure: Mini PCNL — 90 Participants underwent MINI PCNL in MIN PCNL arm and 90 Participants underwent Standard PCNL in Standard PCNL arm.

SUMMARY:
Introduction: Urolithiasis is a common urological condition, and percutaneous nephrolithotomy (PCNL) is a widely used treatment option. Trifecta analysis, which includes stone-free rate, reduced complications (Clavien- Dindo classification), and minimal need for auxiliary procedures, provides a standardized way to compare outcomes. This study evaluates the trifecta outcomes of standard PCNL and mini PCNL.

DETAILED DESCRIPTION:
Methodology: This prospective cohort study was conducted at the department of urology, Institute of Kidney Diseases, Peshawar from Jan 2022 to March 2024. 180 consecutive individuals who were subjected to percutaneous nephrolithotomy (PCNL) were registered for the study. Patients were randomly assigned into two equal groups using a lottery method. Both the standard PCNL group and mini PCNL group consisted of 90 patients each. Patients who required a change in the planned surgical procedure were replaced with new participants from the sample frame. A structured proforma was filled out for all preoperative, perioperative, and postoperative variables in administration of trifecta, and the data was analyzed using SPSS. An assessment was done for predictive factors for the trifecta using logistic regression to calculate the odds ratio, confidence interval (CI), and p value.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 16 and 65 years having renal stones exceeding 20 mm in diameter or having a density more than 1000 Hounsfield Units (HU) were included.

Exclusion Criteria:

* Patients with residual stones following prior PCNL or other endourological procedures or active, untreated urinary tract infections or sepsis or patients with deranged coagulation profiles, were excluded

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Stone free rates | up to 4 weeks on post follow up imaging i.e CT KUB without contrast
  This outcome measures that which modality provide better stone free rates. Mini or standard PCNL.
Post operative complications rate | Up to 4 weeks days post operative period
  To find which modality has got lesser number of complications. Mini or standard PCNL
Need of auxiliary Procedures | Up to 4 weeks post operatively
  to find which modality require the need of auxiliary Procedures like ESWL, URS, or Re DJS stenting.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Kidney Disease., Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
As part of our commitment to research transparency and data-sharing practices, we plan to share individual participant data (IPD) obtained from this clinical trial. The purpose of sharing IPD is to enable further research, facilitate meta-analyses, and contribute to scientific advancements that can improve patient care and clinical outcomes.
  Scope of Data to be Shared
  The de-identified individual participant data that will be shared includes:
  Demographic details such as age, sex, and relevant baseline characteristics Clinical and laboratory data collected during the study Outcome measures related to the study objectives Adverse event reports and safety data All shared data will be de-identified to ensure participant confidentiality and privacy in accordance with applicable ethical guidelines and regulatory requirements.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be made publicly available six months after the primary study results are published in a peer-reviewed journal. The dataset will remain accessible for a period of five years from the initial release, after which continued access will be evaluated based on scientific interest and data usage.
Access Criteria: The IPD will be stored in a secure, electronic form with the principal investigator. Researchers interested in accessing the data will be required to submit a request to the principal author via this email: ahaseeb.dr@gmail.com
  Conditions for Data Access Access to the shared data will be granted to qualified researchers affiliated with recognized academic or clinical institutions. Interested researchers must submit a methodologically sound research proposal outlining the objectives and intended use of the data. Approval will be based on scientific merit and alignment with ethical standards.
  Before access is granted, researchers will be required to:
  Sign a Data Use Agreement (DUA) to ensure appropriate use of the dataset Agree to maintain confidentiality and not attempt to re-identify participants Provide a commitment to acknowledge the original study and funding sources in any resulting publications.
URL: https://medium.com/@imdoc95

REFERENCES:
- Available data/document: Clinical Study Report: 10.7759/cureus — https://www.cureus.com/publish/articles/342384-comparison-of-trifecta-analysis-of-standard-versus-mini-percutaneous-nephrolithotomy-in-the-management-of-urolithiasis/preview#!/ — Further information including data sheets will be provided upon request